CLINICAL TRIAL: NCT05531201
Title: Evaluation of the Efficacy of a Coordinated Interprofessional Care Pathway on Disability in Patients With Chronic Low Back Pain and Patients at Risk of Chronic Low Back Pain in Primary Care: a Cluster Randomized Controlled Trial
Brief Title: Evaluation of the Efficacy of a Coordinated Interprofessional Care Pathway on Disability in Patients With Chronic and at Risk of Chronic Low Back Pain in Primary Care
Acronym: EFFIBACK
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CNGE Conseil (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CNGE-2021/01; 2021-A02432-39 (Registry Identifier: IDRCB)
Record Dates: First submitted 2022-08-22; First posted 2022-09-07 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Physical Therapists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Experimental): Trainig of GP and physiotherapist at collaborative coordinated care pathway
  Interventions: Procedure: collaboration general practitioner and physiotherapist
- Control (No Intervention): without modification of the usual follow-up

INTERVENTIONS:
Procedure: collaboration general practitioner and physiotherapist — training general practitioner and physiotherapist
  Arms: Interventional

SUMMARY:
Low back pain is a public health problem with major individual and socio-economic repercussions. In primary care, strong disparities are observed in the management of low back pain patients. While general practitioners (GPs) and physiotherapists appear as two essential first-line caregivers, collaboration between these professionals remains underdeveloped, most often characterized by a lack of consultation or coordination. Systematic increased interprofessional collaboration is likely to improve the results of the care pathway, by optimizing the existing care offer.

ELIGIBILITY:
Inclusion Criteria:

Adult patients between the ages of 18 and 65

* Patients consulting their GP for a first or new eisode of acute low back pain (more than 12 months from the previous one) with a STarT Back screening tool score greater than 3.
* OR low back pain at risk of chronicity (presence of yellow flags, according to the recommendation of the High Health Authority (HAS) of 2019
* OR recurrent low back pain: in the event of recurrence of low back pain within 12 months after the previous episode, then considered to be at risk of chronicity
* OR having chronic low back pain (low back pain for more than 3 months)
* Patients benefiting from the general social security system
* Patients who understand and speak French fluently
* Patients who have given their consent after having received complete information on the protocol

Exclusion Criteria:

* Minor patients
* Pregnant women (declared pregnancy) or immediately postpartum (up to 3 months)
* Patients with "red flags" (serious neurological impairment, cancer, infection, fracture or inflammatory disease), according to the 2019 HAS recommendation
* Patients referred immediately for imaging or specialist advice during the first consultation with the GP (suspicion of underlying pathology)
* Patients with no history of acute low back pain, at low risk of chronicity (STarT Back screening tool score less than or equal to 3)
* Patients with a contraindication to rehabilitation by physiotherapy
* Patients who have already undergone spine surgery
* Patients with cognitive impairment
* Patients whose life expectancy is less than 12 months
* Patients under guardianship or curatorship, under judicial protection or safeguard of justice
* Patients not affiliated to the general social security system
* Patients with difficulties in understanding the French language
* Patients with an inability to give express consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2026-01-20 (Actual); Study Completion 2026-11-13 (Estimated)

PRIMARY OUTCOMES:
Disability at 3 months | 3 months
  Absolute change in overall Oswestry Disability Index (ODI) scale score between 0 and 3 months. Total score ranging from 0 (no functional disability) to 100 (severe functional disability).

SECONDARY OUTCOMES:
Disability at 12 months | 12 months
  Absolute change in overall ODI scale score between 0 and 12 months. Total score ranging from 0 (no functional disability) to 100 (severe functional disability).
Health-related quality of life at 3 months | 3 months
  Absolute change of health-related quality of life by the EuroQol 5 Dimensions scale (EQ-5D) between 0 and 3 months and between 0 and 12 months
Health-related quality of life at 12 months | 12 months
  Absolute change of health-related quality of life by the EuroQol 5 Dimensions scale (EQ-5D) between 0 and 12 months
Evaluation of the course of care: compliance | 12 months
  number (%) of patients having followed the entire course of care
Evaluation of the course of care: number of consultations | 12 months
  total number of consultations with GPs and physiotherapists (PTs)
Evaluation of the course of care: medical imaging | 12 months
  total number of medical imaging related to low back during the follow up
Evaluation of the course of care: total cost | 12 months
  total cost (in euros €) of healthcare pathway in the two groups
Evaluation of effective collaborative practices | 12 months
  qualitative analysis of GP/PT collaboration using semi-structured interviews with professionals

CONTACTS AND LOCATIONS:
Overall Officials: Tan-Trung PHAN, Study Chair — Département Universitaire d'Enseignement et de Recherche en Médecine Générale - Université Paris-Est Créteil, 8 rue du Général Sarrail 94010 Créteil Cedex
Locations (1):
- Maison de Santé Pluriprofessionnelle Universitaire, Fontainebleau, France

IPD SHARING:
Plan to Share IPD: No